CLINICAL TRIAL: NCT03499847
Title: Assessing the Effectiveness of Different Interventions in Increasing the Completion Rates of the Advanced Medical Directive in the Polyclinic Setting in Singapore - A Randomized Controlled Trial
Brief Title: Increasing the Uptake of Advanced Directives in SingHealth Polyclinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Responsible Party: Principal Investigator, Xu Cunzhi, Family Medicine Resident, SingHealth Polyclinics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Polyclinics AMD Intervention
Record Dates: First submitted 2018-04-08; First posted 2018-04-17 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Advanced Medical Directive, a Legal Document Signed in Advance to State Healthcare Preferences

STUDY DESIGN:
Intervention Model Description: 3-arm, randomised control trial
  1. Active Intervention group (n=65) Counselling provided Pamphlet given
  2. Passive Intervention group (n=65) Pamphlet given
  3. Control group (n=65) Neither counselling nor pamphlet given
Who Masked: Outcomes Assessor
Masking Description: subjects will be interviewed over the telephone 6 weeks after initial intervention by a blinded assessor to assess outcomes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Intervention (Active Comparator): subjects will be given a pamphlet about the advanced medical directive, and a standardized face-to-face counselling session will be conducted with their healthcare provider
  Interventions: Behavioral: standardised face-to-face counselling session; Behavioral: advanced medical directive pamphlet
- Passive Intervention (Active Comparator): subjects will be given a pamphlet about the advanced medical directive
  Interventions: Behavioral: advanced medical directive pamphlet
- Control (No Intervention)

INTERVENTIONS:
Behavioral: standardised face-to-face counselling session — the healthcare provider will conduct a standardised face-to-face counselling session guided with subjects guided by a check-list of topics to cover regarding the Advanced Medical Directive.
  Arms: Active Intervention
Behavioral: advanced medical directive pamphlet — A standardised pamphlet containing information about the Advanced Medical Directive produced by the Ministry of Health, Singapore.
  Arms: Active Intervention; Passive Intervention

SUMMARY:
An Advanced Medical Directive (AMD) is a legal document in Singapore that allows one to inform their medical practitioner that they do not want any life-sustaining treatment should they become unconscious and terminally ill where death is imminent. Despite the AMD act being passed in Singapore Parliament in 1996, uptake remains low among the population. Several intervention studies have shown that education and communication can be effective in promoting end-of-life discussion and planning. In this study, we aim to compare the effectiveness of counselling sessions together with pamphlets, versus pamphlets alone, versus current care, in increasing the completion rates of the AMD in the Singapore Polyclinic setting.

DETAILED DESCRIPTION:
An Advanced Medical Directive (AMD) is a legal document in Singapore that allows one to inform their medical practitioner that they do not want any life-sustaining treatment should they become unconscious and terminally ill where death is imminent. It may be completed by any person, of sound mind, aged 21 years and above.The AMD Act was passed in the Singapore Parliament in May 1996.

A cross-sectional, community-based study surveyed 1200 selected households in Singapore. Only 37.9% of the sample population had heard of the AMD prior to the study, though when approached, 60.6% were willing to sign an AMD. As of 2017, less than 25,000 people (0.45%) in Singapore have opted to sign an AMD.

Past studies have shown that end of life discussions reduce stress, anxiety, and depression in surviving relatives. A local study in 2010 revealed a 33% patient-surrogate discrepancy in end-of-life decision making.

There are a lack of intervention studies regarding AMD in Singapore. In this study, we aim to compare the effectiveness of counselling sessions together with pamphlets, versus pamphlets alone, versus current care, in increasing the completion rates of the AMD in the Singapore Polyclinic setting.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40
* Patient who seeks medical consultation at Singhealth Polyclinics (Bedok, Marine Parade, Outram, Tampines)

Exclusion Criteria:

* History of dementia
* History of depression
* Known diagnosis of terminal illness
* Signed Advanced Medical Directive/Advanced Care Plan previously

Ages: 41 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Number of patients who completed the Advanced Medical Directive | 4 months
Number of patient who expressed interest to complete the Advanced Medical Directive | 4 months

SECONDARY OUTCOMES:
Barriers to completion of the Advanced Medical Directive | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Lian Leng Low, MBBS, Principal Investigator — low.lian.leng@singhealth.com.sg
Locations (4):
- Singapore (4):
  - Outram Polyclinic, Singapore
  - Marine Parade Polyclinic, Singapore
  - Bedok Polyclinic, Singapore
  - Tampines Polyclinic, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tay M, Chia SE, Sng J. Knowledge, attitudes and practices of the Advance Medical Directive in a residential estate in Singapore. Ann Acad Med Singap. 2010 Jun;39(6):424-8. PMID 20625616
- [Background] Ramsaroop SD, Reid MC, Adelman RD. Completing an advance directive in the primary care setting: what do we need for success? J Am Geriatr Soc. 2007 Feb;55(2):277-83. doi: 10.1111/j.1532-5415.2007.01065.x. PMID 17302667
- [Background] Azoulay E, Pochard F, Kentish-Barnes N, Chevret S, Aboab J, Adrie C, Annane D, Bleichner G, Bollaert PE, Darmon M, Fassier T, Galliot R, Garrouste-Orgeas M, Goulenok C, Goldgran-Toledano D, Hayon J, Jourdain M, Kaidomar M, Laplace C, Larche J, Liotier J, Papazian L, Poisson C, Reignier J, Saidi F, Schlemmer B; FAMIREA Study Group. Risk of post-traumatic stress symptoms in family members of intensive care unit patients. Am J Respir Crit Care Med. 2005 May 1;171(9):987-94. doi: 10.1164/rccm.200409-1295OC. Epub 2005 Jan 21. PMID 15665319
- [Background] Foo AS, Lee TW, Soh CR. Discrepancies in end-of-life decisions between elderly patients and their named surrogates. Ann Acad Med Singap. 2012 Apr;41(4):141-53. PMID 22635278
- [Background] Houben CHM, Spruit MA, Groenen MTJ, Wouters EFM, Janssen DJA. Efficacy of advance care planning: a systematic review and meta-analysis. J Am Med Dir Assoc. 2014 Jul;15(7):477-489. doi: 10.1016/j.jamda.2014.01.008. Epub 2014 Mar 2. PMID 24598477
- [Background] Tamayo-Velazquez MI, Simon-Lorda P, Villegas-Portero R, Higueras-Callejon C, Garcia-Gutierrez JF, Martinez-Pecino F, Barrio-Cantalejo IM. Interventions to promote the use of advance directives: an overview of systematic reviews. Patient Educ Couns. 2010 Jul;80(1):10-20. doi: 10.1016/j.pec.2009.09.027. Epub 2009 Oct 29. PMID 19879090
- [Derived] Xu C, Yan S, Chee J, Lee EP, Lim HW, Lim SWC, Low LL. Increasing the completion rate of the advance directives in primary care setting - a randomized controlled trial. BMC Fam Pract. 2021 Jun 18;22(1):115. doi: 10.1186/s12875-021-01473-1. PMID 34144695
- See also: Singapore Ministry of Health - Advanced Medical Directives Information — https://www.moh.gov.sg/policies-and-legislation/advance-medical-directive